CLINICAL TRIAL: NCT00848757
Title: Changing Lifestyles for Better Health: A Model Program for Community Health Centers
Brief Title: Changing Lifestyles for Better Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0903004817
Record Dates: First submitted 2009-02-18; First posted 2009-02-20 (Estimated); Results first posted 2022-03-17 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Lifestyle Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Life-Style Counseling (Experimental): Women with pre-diabetes randomized to the ILI will attend an intensive 12-week group program of nutritional education, diet, behavior modification and structured exercise, which is based on the published curriculum from the Diabetes Prevention Program (DPP) "Lifestyle Balance" program, but modified for a group format and to be more culturally and linguistically appropriate for this population.
  Interventions: Behavioral: Intensive Lifestyle Intervention
- Usual Care Control (No Intervention): Women with pre-diabetes randomized to usual care will be offered 30 minute appointments with a medical provider to review their diagnosis, risk for diabetes, and stress the importance of lifestyle changes to prevent diabetes, including weight loss and exercise and setting individual goals for these. Usual care participants will be encouraged to achieve goals equivalent to the ILI group: to reduce their weight by 7%, and to increase their physical activity to approximately 150 minutes moderate intensity exercise per week. They will be offered a consultation with an FHCHC nutritionist to achieve dietary/weight loss objectives. Participants are offered printed educational materials which are language and literacy-appropriate.

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — Women with pre-diabetes randomized to the ILI will attend an intensive 12-week group program of nutritional education, diet, behavior modification and structured exercise, which is based on the published curriculum from the DPP "Lifestyle Balance" program, but modified for a group format and to be more culturally and linguistically appropriate for this population.
  Arms: Intensive Life-Style Counseling

SUMMARY:
The purpose of this research collaboration between Dr. William Tamborlane, Deputy Directory of the Yale Center for Clinical Investigation (YCCI) and Fair Haven Community Health Center's (FHCHC) Diabetes Prevention Team is to determine the efficacy of an intensive life-style intervention (ILI) program that has been developed and implemented at the FHCHC to prevent the development of diabetes.

DETAILED DESCRIPTION:
This project is a clinical outcome study that merges the expertise of a senior Yale clinical investigator, the clinical and translational research resources of YCCI, the clinical and community expertise of the FHCHC Diabetes Team, and the high-need patient population of FHCHC. In addition to determining the efficacy and cost-effectiveness of an ILI for diabetes prevention in an inner-city community health center setting, this project will evaluate the effectiveness of pooling academic expertise with direct clinical services to disadvantaged, at-risk populations.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for this study, the following criteria must be met:

* Subjects must be willing to travel to the clinic for all regularly scheduled study visits, and to the lifestyle intervention program site for the ILI (the John Martinez School).
* Subjects must have had a 2 hour 75 gram Oral Glucose Tolerance Test (OGTT) with fasting glucose between 100 and 126, or 2 hour glucose between 140 and 200 mg/dl in order to participate in this study within the 4 months prior to enrollment.
* Willingness to undergo fasting blood testing: HOMA-IR, fasting lipid profile (including total cholesterol, HDL, LDL cholesterol and triglycerides) at the beginning of the study (if not previously obtained with the OGTT) and repeated at 12 months.
* Subjects must have no medical contraindications to exercise or dieting.

Exclusion Criteria:

* Subjects will be excluded from the study if they have diabetes or other serious medical or psychiatric condition that would preclude participation in the ILI program.
* Subjects will be excluded if they are taking medications that potentially cause significant weight gain or weight loss (including prescription medication, over the counter medication, or herbal supplements)..
* Women who are pregnant or planning to become pregnant will not be enrolled in this study.
* Any behavioral or psychosocial issue that will interfere with the subject's completion of the program, including an eating disorder will prohibit subjects from participating in this study.
* Subjects cannot participate if they have concurrent membership in a comprehensive weight management program.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2009-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fair Haven Community Health Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Lifestyle Intervention (ILI): Women with pre-diabetes randomized to the ILI will attend an intensive 14-week group program of nutritional education, diet, behavior modification and structured exercise, which is based on the published curriculum from the DPP "Lifestyle Balance" program, but modified for a group format and to be more culturally and linguistically appropriate for this population.
  Intensive Lifestyle Intervention: Women with pre-diabetes randomized to the ILI will attend an intensive 14-week group program of nutritional education, diet, behavior modification and structured exercise, which is based on the published curriculum from the DPP "Lifestyle Balance" program, but modified for a group format and to be more culturally and linguistically appropriate for this population.
Period: Overall Study
Arm/Group | Intensive Lifestyle Intervention (ILI) | Usual Care Control
Started | 65 | 65
Completed | 61 | 61
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Lifestyle Intervention (ILI) | Usual Care Control | Total
Number analyzed (Participants) | 61 | 61 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (10.8) | 43.0 (9.7) | 43 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 61 | 122
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 61 | 122

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: The change is weight is reported from baseline to 12 months.
Time Frame: Baseline and 12 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Intensive Lifestyle Intervention (ILI) | Usual Care Control
Number analyzed (Participants) | 61 | 61
kg | -3.8 [-4.6 to -3.0] | 1.4 [.6 to 2.2]

2. Primary Outcome: Change in BMI
Description: The change in BMI is reported from baseline to 12 months.
Time Frame: Baseline and 12 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Intensive Lifestyle Intervention (ILI) | Usual Care Control
Number analyzed (Participants) | 61 | 61
kg/m^2 | -1.6 [-2 to -1.3] | 0.6 [0.2 to 0.9]

3. Primary Outcome: Change in Percent Body Fat
Description: Change in percent body fat is reported from baseline to 12 months. Body composition by body fat analyzer (TBF-300; Tanita,Arlington Heights, IL) was used.
Time Frame: Baseline and 12 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of body fat
Arm/Group | Intensive Lifestyle Intervention (ILI) | Usual Care Control
Number analyzed (Participants) | 61 | 61
percent of body fat | -1.9 [-2.9 to -1.0] | 0.4 [-0.7 to 1.4]

4. Primary Outcome: Change in Waist Circumference
Description: Change in waist circumference was measured from baseline to 12 months
Time Frame: Baseline and 12 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Intensive Lifestyle Intervention (ILI) | Usual Care Control
Number analyzed (Participants) | 61 | 61
cm | -3.3 [-5.2 to -1.4] | -0.2 [-2.1 to 1.7]

5. Primary Outcome: Change in Blood Pressure
Description: Change in blood pressure was measured from baseline to 12 months
Time Frame: Baseline and 12 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Intensive Lifestyle Intervention (ILI) | Usual Care Control
Number analyzed (Participants) | 61 | 61
mm Hg
  Systolic blood pressure | -1.5 [-5.0 to 2.1] | 0 [-3.6 to 3.6]
  Diastolic blood pressure | -0.5 [-2.8 to 1.7] | -0.9 [-3.2 to 1.4]

6. Secondary Outcome: Physical Activity Levels (Self-reported)
Time Frame: 12 months
Population: Data was not collected.
Arm/Group | Intensive Lifestyle Intervention (ILI) | Usual Care Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Usual Care Control | Intensive Lifestyle Intervention (ILI)
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No